CLINICAL TRIAL: NCT03572699
Title: Simple, Mobile-based Artificial Intelligence AlgoRithms in the Detection of Diabetic ReTinopathy (SMART) Study
Acronym: SMART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medios Technologies Pte. Ltd (Industry)
Collaborators: Diacon Hospital (Other)
Responsible Party: Principal Investigator, Dr Srikanth Y N, Principal investigator, Medios Technologies Pte. Ltd
Other Study IDs: SMART1
Record Dates: First submitted 2018-06-16; First posted 2018-06-28 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: diabetic retinopathy — This is an observational study of patients with diabetes. Patients undergoing routine care will undergo retinal imaging using a nonmydriatic fundus camera. The images will be run on an artificial intelligence (AI) algorithm. The diagnosis of the artificial intelligence algorithm will be compared to the image diagnosis given by the ophthalmologists. The ophthalmologists will be blinded to the diagnosis of the AI and vice versa. The data will be analyzed to evaluate the performance of the AI.

SUMMARY:
This is an observational cross sectional study aimed to evaluate the performance of the artificial intelligence algorithm in detecting any grade of diabetic retinopathy using retinal images from patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 1 or type 2 diabetes mellitus
2. Ages 18 and above
3. Male and female

Exclusion Criteria:

1. Persistent visual impairment in one or both eyes;
2. Subjects with corneal opacities and advanced cataract.
3. History of retinal vascular (vein or artery) occlusion;
4. Subject is contraindicated for fundus photography (for example, has light sensitivity);
5. Subject is currently enrolled in an interventional study of an investigational device or drug;
6. Subject has a condition or is in a situation which in the opinion of the Investigator, might confound study results, may interfere significantly with the subject's participation in the study, or may result in ungradable clinical reference standard photographs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with diabetes mellitus presenting to the outpatient for routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2018-07-11 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the AI in detecting any grade of diabetic retinopathy | 3 months

SECONDARY OUTCOMES:
Sensitivity and specificity of the AI in detecting referable diabetic retinopathy (referable retinopathy defined as moderate non proliferative retinopathy or greater) | 3 months
Sensitivity and specificity of the AI in detecting sight threatening diabetic retinopathy (referable retinopathy defined as severe non proliferative retinopathy or greater) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Srikanth Y N, MS, Principal Investigator — Investigator
Locations (1):
- Diacon Hospital, Bangalore, India

IPD SHARING:
Plan to Share IPD: No